CLINICAL TRIAL: NCT00337155
Title: A Double Blind, Randomised, Dose Finding, Repeat Dose, Phase II, Multicentre Study of Alpharadin® for the Treatment of Patients With Hormone Refractory Prostate Cancer and Skeletal Metastases
Brief Title: BAY88-8223, Dose Finding Study in Patients With HRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15304; 2005-003680-22 (EudraCT Number); BC1-04 (Other: Algeta ASA)
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2014-12

CONDITIONS: Prostate Cancer; Neoplasm Metastasis
Keywords: Recurrent Prostate Cancer; metastatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Radium-223 dichloride (Xofigo, BAY88-8223) Dose group 1 (Experimental): 25 kBq/kg b.w., 3 times at 6 week intervals
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)
- Radium-223 dichloride (Xofigo, BAY88-8223) Dose group 2 (Experimental): 50 kBq/kg b.w., 3 times at 6 week intervals
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)
- Radium-223 dichloride (Xofigo, BAY88-8223) Dose group 3 (Experimental): 80 kBq/kg b.w., 3 times at 6 week intervals
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (BAY88-8223) — 3 doses of radium-223 at different dose levels, 25, 50 or 80 kBq/kg b.w.given as injection.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the investigational radioisotope Radium-223, Alpharadin, in treatment of men with prostate cancer and bone metastases that no longer respond to hormonal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Hormone refractory with evidence of rising PSA:

  * Patient must be maintained on androgen ablation therapy with LHRH agonist (stable dose for at least 8 weeks prior to study entry), or have undergone orchiectomy
  * Serum testosterone level is required to be ≤ 50 ng/dl
  * Patients who have received prior hormonal drug therapy:

    * Flutamide, nilutamide or cyproterone acetate must have stopped at least four weeks prior to study drug administration and progression must have been demonstrated since cessation;
    * Bicalutamide must have stopped at least six weeks prior to study drug administration and progression must have been demonstrated since cessation
  * Elevated and rising PSA:

    * Baseline PSA level ≥ 10 ng/ml
    * Progressive rise in PSA, defined as two consecutive increases in PSA documented over a previous reference value (measure 1). The first increase in PSA (measure 2) should occur a minimum of 1 week from the reference value (measure 1. This increase in PSA should be confirmed (measure 3) after a minimum of 1 week. If the confirmatory PSA value (measure 3) is less than the previous value, the patient will still be eligible provided the next PSA measure (measure 4)is found to be greater than the second PSA value(measure 2).3. Multifocal skeletal metastases confirmed by bone scintigraphy within the last 6 weeks
* Performance status: ECOG 0-2
* Life expectancy: At least 6 months
* Laboratory requirements:

  * Neutrophil count ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x109/L
  * Haemoglobin ≥ 95 g/L
  * Total bilirubin level within normal institutional limits
  * ASAT and ALAT ≤ 2,5 times upper institutional limit of the normal range
* The patient is willing and able to comply with the protocol (including maintenance of patient diary), and agrees to return to the hospital for follow-up visits and examination
* The patient has been fully informed about the study and has signed the informed consent form

Exclusion Criteria:

* Has received an investigational drug within 4 weeks prior to the administration of radium-223, or is scheduled to receive one during the treatment and post-treatment period
* Has received chemo-, immunotherapy, or external radiotherapy within the last 4 weeks prior to administration of study drug, or has not recovered from adverse events due to agents administered more than 4 weeks earlier
* More than one regimen of previous cytotoxic chemotherapy
* Has received prior hemibody external radiotherapy
* Has a need for immediate external radiotherapy
* Has received systemic radiotherapy with strontium-89, samarium-153, rhenium-186 or rhenium-188 for the treatment of bony metastases within the last year prior to administration of study drug
* Has started treatment with bisphosphonates less than 3 months prior to administration of study drug. Patients are allowed to be on bisphosphonates provided patient is on a stable dose for ≥ 12 weeks before administration of study drug.
* Patients who are ≤ 4 weeks (6 weeks for bicalutamide) post withdrawal of antiandrogen therapy
* Patients who have started or stopped systemic steroids, within a week prior to study drug administration
* Other currently active (relapse within the last 3 years) malignancy (except non-melanoma skin cancer) that are not prostate cancer metastases
* Visceral metastases from prostate cancer as assessed by abdominal/pelvic CT or MRI within six weeks before administration of study drug; Lung lesions from prostate cancer as assessed by chest X-ray within 6 weeks. This requirement does not include abdominal or pelvic lymph node involvement (individual lymph node size must not exceed 1 cm in short diameter) which is acceptable
* Bulky loco-regional disease
* Any other serious illness or medical condition, for example:

  * any uncontrolled infection
  * any patient who has clinical heart failure severe enough to cause marked limitation of activity, and who is only comfortable at rest; or any patient who has heart failure more severe than this (NYHA Heart Failure Class III or IV
  * Crohns disease or ulcerative colitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants in each dose group with a confirmed PSA response | 24 weeks, 12 months, 24 months
  PSA response; each patient will be classified as PSA responder/non-responder according to the definition of PSA response:a decrease from baseline of at least 50% maintained for at least three weeks.

SECONDARY OUTCOMES:
The maximum percent decrease in PSA level compared to baseline | 24 weeks, 12 months, 24 months
Time to PSA Progression | 24 weeks, 12 months, 24 months
Bone-ALP response (classified as for PSA response) and decrease in bone-ALP level compared to baseline | 24 weeks, 12 months, 24 months
Total number of SRE per patient | 24 weeks, 12 months, 24months
Pain Assessment and analgesic consumption | 24 weeks, 12 months, 24months
Time to death from first treatment | 24 weeks, 12 months, 24months
Time to Skeletal Related Events (SRE) | 24 weeks, 12 months, 24 months
Adverse events, blood chemistry and haematological toxicity | 24 weeks, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Sutton, Surrey, United Kingdom

REFERENCES:
- [Result] Parker CC, Pascoe S, Chodacki A, O'Sullivan JM, Germa JR, O'Bryan-Tear CG, Haider T, Hoskin P. A randomized, double-blind, dose-finding, multicenter, phase 2 study of radium chloride (Ra 223) in patients with bone metastases and castration-resistant prostate cancer. Eur Urol. 2013 Feb;63(2):189-97. doi: 10.1016/j.eururo.2012.09.008. Epub 2012 Sep 13. PMID 23000088